CLINICAL TRIAL: NCT01540968
Title: Influence of a Combined Intervention by Nutritional Support and Physical Exercise on Quality of Life in Cancer Out-patients Treated in Palliative Intention.
Brief Title: Nutrition and Physical Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KEK-ZH-Nr. 2011-0447; KFS-2833-08-2011 (Other Grant/Funding Number: Krebsforschung Schweiz / Krebsliga Schweiz)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Gastrointestinal Cancer; Lung Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition & physical exercise (Experimental)
  Interventions: Behavioral: Nutrition & physical exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Nutrition & physical exercise — Patients will be randomly assigned to intensive individual nutritional counselling including oral nutritional supplements and a specifically designed exercise program combining strength and balance training.
  Arms: Nutrition & physical exercise

SUMMARY:
The purpose of this study is to investigate the effect of a combined treatment of nutritional therapy and physical exercise in palliative cancer out-patients. The investigators hypothesize that this combined intervention consisting of an increased energy- and protein intake and physical exercise level improves quality of life (QoL), functional and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic lung cancer or gastrointestinal cancer
* WHO performance status 0, 1 or 2
* Able to walk at least 100 meters independently without crutches or walking frame assessed by the treating physician on the basis of the patient's history and physical condition
* Receiving palliative treatment

Exclusion Criteria:

* Enteral and/or parenteral nutrition within 1 month previous to study participation
* History of ileus within one month
* Known brain metastases or symptomatic bone metastases
* Psychiatric disorder precluding understanding of information on trial related topics and giving informed consent.
* Any serious underlying medical condition which could impair the ability of the patient to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Ballmer, Prof. Dr., Study Chair — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland